CLINICAL TRIAL: NCT06018675
Title: Comparison of Kinesio Taping, Dry Needling and Lidocain Injection Methods in Myofascial Pain Syndrome
Status: Completed | Type: Observational
Sponsor: Bursa City Hospital (Other Government)
Responsible Party: Principal Investigator, Sezin Solum, MD; Physical Medicine & Rehabilitation Specialist Physician, Bursa City Hospital
Other Study IDs: 9999999993
Record Dates: First submitted 2023-08-22; First posted 2023-08-31 (Actual); Last update posted 2023-08-31 (Actual); Status verified 2023-08

CONDITIONS: Myofascial Pain Syndrome
Keywords: myofascial pain syndrome; dry needling; kinesiotherapy; lidocain injection; quality of life
MeSH Terms: conditions — Myofascial Pain Syndromes | interventions — Dry Needling

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Group 1: Kinesiotherapy
  Interventions: Other: kinesiotherapy
- Group 2: Dry needling
- Group 3: Lidocain injection

INTERVENTIONS:
Other: kinesiotherapy — Group 1: Kinesiotherapy Group 2: Dry needling Group 3: lidocain injection
  Other Names: dry needling; lidocain injection
  Groups: Group 1

SUMMARY:
Myofascial pain syndrome (MPS) is a chronic pain syndrome characterized by the presence of trigger points in muscles and fascia in various parts of the body. Due to the pain, it has negative effects on function, restricting movements and daily life activities. Several invasive and non-invasive methods with proven effectiveness are described in the management of myofascial pain syndrome. In this study, investigators aimed to compare the effect of kinesiotaping with dry needling and lidocaine injection treatment. İnvestigators hypothesized, that the effect of kinesiotaping have similar results compared to the invasiv treatment methods in the treatment of MPS.

Sixty-six patients diagnosed with myofascial pain syndrome in the upper trapezius were included in this retrospective study. Patients were divided into three groups. Twenty-two patients were randomly selected among patients who received kinesiotaping treatment (n:22). Twenty-two patients who received dry needling treatment (group 2) and 22 patients who received lidocaine injection treatment were randomly selected as controls. Patients were evaluated using the Visual Analogue Scale (VAS) and the Short Form (SF-36) scales, which were completed before and 3 weeks after the treatment.

DETAILED DESCRIPTION:
Myofascial pain syndrome (MPS) is a chronic pain syndrome characterized by the presence of trigger points in muscles and fascia in various parts of the body. Myofascial pain syndrome is one of the most common musculoskeletal problems in adults, and its prevalence varies between 30-93%. Patients have symptoms such as pain (local or referred), loss of muscle strength, stiffness, and restriction of range of motion. Although the etiology of myofascial pain syndrome is not well understood, causes such as posture disorder, trauma, and ergonomic problems appear as etiology. Simon criteria are often used in the diagnosis. Apart from this, anamnesis and detailed physical examination are important in the diagnosis of MPS.

Dry needling is a treatment method which uses needles similar to those used in acupuncture, without any injectable drug to myofascial trigger points. Dry needling shows its effect through the exposure to various chemical mediators. The observation of a local course response in dry needling shows that the treatment is effective. Side effects such as bleeding, localized pain, vasovagal syncope, and rarely pneumothorax may occur during the treatment of dry needling.

Lidocaine injection and Dry needling are different applications that injectable drugs are not use in dry needling. Lidocain injection applied by giving a local anesthetic substance on the trigger point. It has been reported in the conducted studies that it has a similar effect as dry needling and that local pain is less common after injection.

Kinesiotaping (KT) is a treatment method developed by Dr. Kenzo Kase, which has been initially applied in the treatment of pain, and its use has become widespread in recent years. KT tape is a thin and flexible tape that allows joint movements. KT tape is widely used in the treatment of pain relief, muscle relaxation, edema reducement, improvement of muscle strength, and posture correction. Although the exact mechanism of KT is not well known, it is believed to cause a decrease in nociceptor pressure, create a space in the subcutaneous area, convenience in the removal of chemical mediators from the tissue, and also stimulation of somotosensory and proprioceptive mechanisms.

In our study, investigators aimed to compare the effectiveness of non-invasive KT on myofascial pain syndrome treatment with invasive treatment methods such as dry needling and lidocaine injections. The investigators hypothesized, that the effect of kinesiotherapy have similar results compared to the invasiv treatment methods in the management of MPS.

After IRB approval and informed consent by all patients were obtained, investigators performed this retrospective study. Instutional review board was obtained by the ethics committee of Bağcılar Training and Research Hospital (Number: 018.07.2.03.057.r1.071). All patients between 18-70 years who were diagnosed with myofascial pain syndrome in the upper trapezius muscle between January 2017 to December 2018 at investigator 's institution were enrolled in this study. According to the power analysis result, 22 patients files were randomly selected among the patients received KT (group 1) using the coin method, and 22 files were randomly selected from the files of patients receiving dry needling (group 2) and lidocaine injection (group 3) treatment in the same way. There were no differences between the age and gender distributions of all 3 selected groups. Patients, who have received conventional physical therapy in the last 6 months, diagnosed with fibromyalgia or fibromyalgia treatment, with a history of neurological disease, malignancy, cervical disc hernia, and who have undergone surgical intervention in the shoulder or neck region or who have received treatment for the diagnosis of myofascial pain syndrome in the last year were excluded from our study.

All 3 treatment modalities were applied to the patients by the same physician. KT treatment was performed using the pain inhibition technique for KT treatment recipients in group 1 (n=22). A total of 3 sessions, one week apart, were applied to the patients using the application of KinesioTex Gold Band. Patients received the treatment in a sitting position. The application was performed while the patients were in the sitting position with the neck in lateral flexion and rotation to the contralateral side. Two 15 cm and 20 cm bands were used in the application, respectively. The first band origin was adhered to the acromion, maximum tension was applied to the first 5-6 cm of tape. Tension was not applied to the rest of the band. The second band was cut in a Y-shape. The application's origin was acromion. The upper part of the Y legs of the tape was applied to the C7 spinosus process and the lower part was applied to the T12 region. Maximum stress was applied to both ends of the tape.

The patients in group 2 who underwent dry needling were applied with 0.25x25 mm sterile acupuncture needles after cleaning the skin with alcohol while in a sitting position. The pistoning was performed on the trigger points in a radial manner and until the local twitch response was obtained. The needles were left in the pistoning area for another 10 minutes after the twitch response was obtained.

The pistoning was made to the patients in Group 3, sitting in an upright position. 2% lidocaine was injected with 26 Gauchl 0.45x13 mm disposable sterile needles into 3 trigger points where the pain was most felt, after sterilizing the skin with a local antiseptic.

All three groups underwent trapeze stretching exercises and were not given any medical treatment.

All patients were evaluated with VAS and SF-36 form before and 3 weeks after treatment. The VAS scale is a pain scale with marked 0-10 areas. Zero represents the absence of pain, while 10 represents very severe pain. The SF-36 form consists of 36 items to evaluate the daily life activities of the patients. It is used to evaluate many daily life functions such as general health status, physical condition, social status, emotional state. A high SF-36 score is one of the indicators of well-being in health.

ELIGIBILITY:
Inclusion Criteria:

* Beetween the age of 18-70
* Presence of myofascial pain syndrome in the upper trapezius muscle

Exclusion Criteria:

* Received conventional physical therapy in the last 6 months
* Diagnosed with fibromyalgia or fibromyalgia treatment
* History of neurological disease, malignancy, cervical disc hernia
* Undergone surgical intervention in the shoulder or neck region
* Received treatment for the diagnosis of myofascial pain syndrome in the last year

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients between 18-70 years who were diagnosed with myofascial pain syndrome in the upper trapezius muscle between January 2017 to December 2018 at our institution were enrolled in this study. According to the power analysis result, 22 patients files were randomly selected among the patients received KT (group 1) using the coin method, and 22 files were randomly selected from the files of patients receiving dry needling (group 2) and lidocaine injection (group 3) treatment in the same way.
Sampling Method: Probability Sample
Enrollment: 66 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2019-01-01 (Actual); Study Completion 2019-08-01 (Actual)

PRIMARY OUTCOMES:
Visual Analog Scala (VAS) | All patients were evaluated with VAS and SF-36 form before and 3 weeks after treatment.
  The VAS scale is a pain scale with marked 0-10 areas. Zero represents the absence of pain, while 10 represents very severe pain.
Short form-36 (SF-36) | All patients were evaluated with VAS and SF-36 form before and 3 weeks after treatment.
  The SF-36 form consists of 36 items to evaluate the daily life activities of the patients. It is used to evaluate many daily life functions such as general health status, physical condition, social status, emotional state. A high SF-36 score is one of the indicators of well-being in health.

CONTACTS AND LOCATIONS:
Overall Officials: Seher Kara, MD, Study Director — Gaziosmapaşa Training and Research Hospital

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Dogan N, Sengul I, Akcay-Yalbuzdag S, Kaya T. Kinesio taping versus dry needling in the treatment of myofascial pain of the upper trapezius muscle: A randomized, single blind (evaluator), prospective study. J Back Musculoskelet Rehabil. 2019;32(5):819-827. doi: 10.3233/BMR-181162. PMID 30883331
- [Background] Ay S, Konak HE, Evcik D, Kibar S. The effectiveness of Kinesio Taping on pain and disability in cervical myofascial pain syndrome. Rev Bras Reumatol Engl Ed. 2017 Mar-Apr;57(2):93-99. doi: 10.1016/j.rbre.2016.03.012. Epub 2016 May 10. English, Portuguese. PMID 28343625
- [Background] Albagieh H, Aloyouny A, Alshehri N, Alsammahi N, Almutrafi D, Hadlaq E. Efficacy of lidocaine versus mepivacaine in the management of myofascial pain. Saudi Pharm J. 2020 Oct;28(10):1238-1242. doi: 10.1016/j.jsps.2020.08.014. Epub 2020 Aug 28. PMID 33132718
- [Background] Raeissadat SA, Rayegani SM, Sadeghi F, Rahimi-Dehgolan S. Comparison of ozone and lidocaine injection efficacy vs dry needling in myofascial pain syndrome patients. J Pain Res. 2018 Jun 29;11:1273-1279. doi: 10.2147/JPR.S164629. eCollection 2018. PMID 29988746
- [Background] Kalichman L, Vulfsons S. Dry needling in the management of musculoskeletal pain. J Am Board Fam Med. 2010 Sep-Oct;23(5):640-6. doi: 10.3122/jabfm.2010.05.090296. PMID 20823359
- [Background] Gerber LH, Shah J, Rosenberger W, Armstrong K, Turo D, Otto P, Heimur J, Thaker N, Sikdar S. Dry Needling Alters Trigger Points in the Upper Trapezius Muscle and Reduces Pain in Subjects With Chronic Myofascial Pain. PM R. 2015 Jul;7(7):711-718. doi: 10.1016/j.pmrj.2015.01.020. Epub 2015 Feb 4. PMID 25661462
- [Background] Ghasemi M, Mosaffa F, Hoseini B, Behnaz F. Comparison of the Effect of Bicarbonate, Hyaluronidase, and Lidocaine Injection on Myofascial Pain Syndrome. Anesth Pain Med. 2020 Jun 23;10(3):e101037. doi: 10.5812/aapm.101037. eCollection 2020 Jun. PMID 32944559
- [Background] Fricton J. Myofascial Pain: Mechanisms to Management. Oral Maxillofac Surg Clin North Am. 2016 Aug;28(3):289-311. doi: 10.1016/j.coms.2016.03.010. PMID 27475508
- [Background] Shah JP, Thaker N, Heimur J, Aredo JV, Sikdar S, Gerber L. Myofascial Trigger Points Then and Now: A Historical and Scientific Perspective. PM R. 2015 Jul;7(7):746-761. doi: 10.1016/j.pmrj.2015.01.024. Epub 2015 Feb 24. PMID 25724849
- [Background] Fleckenstein J, Zaps D, Ruger LJ, Lehmeyer L, Freiberg F, Lang PM, Irnich D. Discrepancy between prevalence and perceived effectiveness of treatment methods in myofascial pain syndrome: results of a cross-sectional, nationwide survey. BMC Musculoskelet Disord. 2010 Feb 11;11:32. doi: 10.1186/1471-2474-11-32. PMID 20149248
- [Background] Onat SS, Polat CS, Bicer S, Sahin Z, Tasoglu O. Effect of Dry Needling Injection and Kinesiotaping on Pain and Quality of Life in Patients with Mechanical Neck Pain. Pain Physician. 2019 Nov;22(6):583-589. PMID 31775405
- [Background] Ozturk G, Kulcu DG, Mesci N, Silte AD, Aydog E. Efficacy of kinesio tape application on pain and muscle strength in patients with myofascial pain syndrome: a placebo-controlled trial. J Phys Ther Sci. 2016 Apr;28(4):1074-9. doi: 10.1589/jpts.28.1074. Epub 2016 Apr 28. PMID 27190430
- [Background] Yilmaz N, Erdal A, Demir O. A comparison of dry needling and kinesiotaping therapies in myofascial pain syndrome: A randomized clinical study. Turk J Phys Med Rehabil. 2020 Aug 18;66(3):351-359. doi: 10.5606/tftrd.2020.3917. eCollection 2020 Sep. PMID 33089092
- [Background] Noguera-Iturbe Y, Martinez-Gramage J, Montanez-Aguilera FJ, Casana J, Lison JF. Short-Term Effects of Kinesio Taping in the Treatment of Latent and Active Upper Trapezius Trigger Points: two Prospective, Randomized, Sham-Controlled Trials. Sci Rep. 2019 Oct 9;9(1):14478. doi: 10.1038/s41598-019-51146-4. PMID 31597934